CLINICAL TRIAL: NCT02498353
Title: Preoperative Short-course Radiotherapy With Local Boost Versus Conventional Preoperative Short-course Radiotherapy for Rectal Cancer
Brief Title: Comparing Preoperative Short-course Radiotherapy With or Without Local Boost for Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Zhou Fuxiang, professor, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZNHCR
Record Dates: First submitted 2015-06-28; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): Preoperative short-course radiotherapy with local boost ,the dose of radiotherapy is PTV-CTV 25Gy/5F with local boost of PTV-GTV 30Gy/5F.
  TME surgery after radiotherapy.
  Interventions: Radiation: preoperative short-course radiotherapy with local boost; Procedure: TME surgery
- control group (Active Comparator): Preoperative short-course radiotherapy without local boost,the dose of radiotherapy is PTV-CTV 25Gy/5F without local boost.
  TME surgery after radiotherapy.
  Interventions: Radiation: preoperative short-course radiotherapy without local boost; Procedure: TME surgery

INTERVENTIONS:
Radiation: preoperative short-course radiotherapy with local boost — Except the clinical target volume(CTV),a gross tumour volume（GTV）is delineated，and give a dose of PTV-GTV:30Gy/5F
  Arms: study group
Radiation: preoperative short-course radiotherapy without local boost — Preoperative short-course radiotherapy without local boost,the dose of radiotherapy is PTV-CTV 25Gy/5F
  Arms: control group
Procedure: TME surgery — both study group and control group received surgery under TME principle after radiotherapy

SUMMARY:
A randomized trial comparing weather preoperative short-course radiotherapy with local boost is better than conventional preoperative short-course radiotherapy for local advanced rectal cancer.

DETAILED DESCRIPTION:
The study plans to recruit 100 patients,randomized into study group and control group,patients in study group are given the dose of PTV(planned target volume)-CTV(clinical target volume) 25Gy/5F with a local boost of PTV-GTV(gross tumour volume) 30Gy/5F；patients in control group are given the dose of PTV-CTV 25Gy/5F without a local boost. The other inventions are the same during the whole treatment,after the radiotherapy,they will receive a surgery under TME((total mesorectal excision) principal.Comparing the toxicity of radiotherapy, R0 resection rate,pathological complete remission rate, complications of operation and sphincter retention rate of these two groups to find out weather local boost bringing benefits to patients with local advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Local advanced rectal cancer (TNM Stage ：T3-4NxM0 )diagnosed by biopsy and MRI or Endoscopic ultrasonography .
* distance between tumour and anal edge ≤12cm.
* PS（(Performance Status） score 0-2 or Karnofsky score≥70.
* liver and kidney functions are normal.
* without any treatment before inclusion.

Exclusion Criteria:

* metastasis
* combined with other severe diseases，such as other kind of cancer ,COPD,myocardial infarction,ect.
* include in other clinical trails.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
pathological complete remission rate | 4 weeks after the surgery

SECONDARY OUTCOMES:
disease free survival | From date of randomization until the date of first documented progression，assessed up to 60 months
sphincter retention rate | 4 weeks after the surgery
toxicity of radiotherapy based on the CTCAE v3.0 (common terminology criteria for adverse events，CTCAE v3.0) | up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Fuxiang Zhou, professor, Study Director — Zhongnan Hospital

REFERENCES:
- [Result] Inra JA, Syngal S. Colorectal cancer in young adults. Dig Dis Sci. 2015 Mar;60(3):722-33. doi: 10.1007/s10620-014-3464-0. Epub 2014 Dec 6. PMID 25480403
- [Result] Sauer R, Fietkau R, Wittekind C, Rodel C, Martus P, Hohenberger W, Tschmelitsch J, Sabitzer H, Karstens JH, Becker H, Hess C, Raab R; German Rectal Cancer Group. Adjuvant vs. neoadjuvant radiochemotherapy for locally advanced rectal cancer: the German trial CAO/ARO/AIO-94. Colorectal Dis. 2003 Sep;5(5):406-15. doi: 10.1046/j.1463-1318.2003.00509.x. PMID 12925071
- [Result] Sauer R, Liersch T, Merkel S, Fietkau R, Hohenberger W, Hess C, Becker H, Raab HR, Villanueva MT, Witzigmann H, Wittekind C, Beissbarth T, Rodel C. Preoperative versus postoperative chemoradiotherapy for locally advanced rectal cancer: results of the German CAO/ARO/AIO-94 randomized phase III trial after a median follow-up of 11 years. J Clin Oncol. 2012 Jun 1;30(16):1926-33. doi: 10.1200/JCO.2011.40.1836. Epub 2012 Apr 23. PMID 22529255
- [Result] Folkesson J, Birgisson H, Pahlman L, Cedermark B, Glimelius B, Gunnarsson U. Swedish Rectal Cancer Trial: long lasting benefits from radiotherapy on survival and local recurrence rate. J Clin Oncol. 2005 Aug 20;23(24):5644-50. doi: 10.1200/JCO.2005.08.144. PMID 16110023
- [Result] Guckenberger M, Saur G, Wehner D, Thalheimer A, Kim M, Germer CT, Flentje M. Long-term quality-of-life after neoadjuvant short-course radiotherapy and long-course radiochemotherapy for locally advanced rectal cancer. Radiother Oncol. 2013 Aug;108(2):326-30. doi: 10.1016/j.radonc.2013.08.022. Epub 2013 Sep 7. PMID 24021342
- [Result] Peeters KC, Marijnen CA, Nagtegaal ID, Kranenbarg EK, Putter H, Wiggers T, Rutten H, Pahlman L, Glimelius B, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. The TME trial after a median follow-up of 6 years: increased local control but no survival benefit in irradiated patients with resectable rectal carcinoma. Ann Surg. 2007 Nov;246(5):693-701. doi: 10.1097/01.sla.0000257358.56863.ce. PMID 17968156
- [Result] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Result] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Result] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Result] Ngan SY, Burmeister B, Fisher RJ, Solomon M, Goldstein D, Joseph D, Ackland SP, Schache D, McClure B, McLachlan SA, McKendrick J, Leong T, Hartopeanu C, Zalcberg J, Mackay J. Randomized trial of short-course radiotherapy versus long-course chemoradiation comparing rates of local recurrence in patients with T3 rectal cancer: Trans-Tasman Radiation Oncology Group trial 01.04. J Clin Oncol. 2012 Nov 1;30(31):3827-33. doi: 10.1200/JCO.2012.42.9597. Epub 2012 Sep 24. PMID 23008301
- [Result] Ortholan C, Romestaing P, Chapet O, Gerard JP. Correlation in rectal cancer between clinical tumor response after neoadjuvant radiotherapy and sphincter or organ preservation: 10-year results of the Lyon R 96-02 randomized trial. Int J Radiat Oncol Biol Phys. 2012 Jun 1;83(2):e165-71. doi: 10.1016/j.ijrobp.2011.12.002. PMID 22579379
- [Result] Faria S, Kopek N, Hijal T, Liberman S, Charlebois P, Stein B, Meterissian S, Meguerditchian A, Fawaz Z, Artho G. Phase II trial of short-course radiotherapy followed by delayed surgery for locoregionally advanced rectal cancer. Colorectal Dis. 2014 Feb;16(2):O66-70. doi: 10.1111/codi.12466. PMID 24148225
- [Result] Bujko K, Partycki M, Pietrzak L. Neoadjuvant radiotherapy (5 x 5 Gy): immediate versus delayed surgery. Recent Results Cancer Res. 2014;203:171-87. doi: 10.1007/978-3-319-08060-4_12. PMID 25103005